CLINICAL TRIAL: NCT01680718
Title: Neuropeptides and Social Behavior
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Naomi Eisenberger, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: Behavioral Neuropeptides
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Social Psychology
Keywords: oxytocin; vasopressin; intranasal administration; healthy sample
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intranasal oxytocin (Experimental): Participants will self-administer 24 IU oxytocin (Syntocinon, Novartis Pharmaceuticals). 5 puffs per nostril (1 puff = 2.4 IU oxytocin).
  Interventions: Drug: Intranasal oxytocin
- Intranasal vasopressin (Experimental): Participants will self-administer 20 IU vasopressin (American Regent Pharmaceuticals). 5 puffs per nostril (1 puff = 2 IU vasopressin).
  Interventions: Drug: Intranasal vasopressin
- Intranasal placebo (Placebo Comparator): 2 mls Glycerine and 3 mls purified water (methylparaben and propylparaben mixed according to purified water formula) for a total of 5 ml, which will be filtered with a 5mu filter (used previously; Bartz et al., 2010). Participants will self-administer 5 puffs per nostril.
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — Through the use of 1oz bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 24 IU oxytocin (Syntocinon, Novartis Pharmaceuticals). 5 puffs per nostril (1 puff = 2.4 IU oxytocin).
  Other Names: Syntocinon nasal spray
  Arms: Intranasal oxytocin
Drug: Intranasal vasopressin — Through the use of 1oz bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 20 IU vasopressin (American Regent Pharmaceuticals). 5 puffs per nostril (1 puff = 2 IU vasopressin).
  Arms: Intranasal vasopressin
Drug: Intranasal placebo — Through the use of 1oz bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 5 puffs per nostril. Placebo consists of: 2 mls Glycerine and 3 mls purified water (methylparaben and propylparaben mixed according to purified water formula) for a total of 5 ml, which will be filtered with a 5mu filter (used previously; Bartz et al., 2010).
  Arms: Intranasal placebo

SUMMARY:
It has long been established that interpersonal relationships can have a profound impact on health and well-being. Yet, we are still learning about the complex biological processes that contribute to positive social interactions and the ability to develop and maintain social relationships. Recent research has begun to focus on oxytocin and vasopressin, neuropeptides that are naturally produced in the hypothalamus, because administration of these neuropeptides has been associated with increased trust, generosity, empathy, cooperation, memory of social stimuli (e.g., faces), and brain activity in neural regions associated with social and emotional processes. To date, several aspects of oxytocin and vasopressin's effects on social behavior have been unexplored. As such, the overarching goal of this project is to examine the effects of intranasal oxytocin and vasopressin on social working memory, deception detection, sensitivity to interpersonal distance, empathy, and altruistic behavior. Understanding how oxytocin and vasopressin influence these aspects of social functioning will help to inform research that has begun to establish the potential for use of these neuropeptides in psychiatric disorders such as autism spectrum disorders and schizophrenia that are characterized by social deficits. For this study, we will recruit 150 healthy adults without a history of medical or psychiatric illness to come to the laboratory. In the first session, participants will complete several questionnaires. In the second session, participants will be randomly assigned to receive oxytocin, vasopressin, or placebo. The study nurses will measure temperature, heart rate, and blood pressure (female participants will also be asked to undergo a pregnancy test) before drug administration. Participants will then complete computer tasks. During the second session, we will also collect a saliva sample for genetic analysis and participants will be asked to complete several additional questionnaires. At the end of the experimental session, participants will be fully debriefed.

The investigators hypothesize that compared to placebo, oxytocin and/or vasopressin will improve social working memory and deception detection, and increase empathy and altruism. It is also hypothesized that main effects will not be found for oxytocin or vasopressin, but rather, analyses of relevant moderators will elucidate these findings.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Healthy (see below)
* Fluent in English

Exclusion Criteria:

* Women who gave birth in the last six months, are currently pregnant, planning to become pregnant in the next 6 months, or currently breastfeeding women
* Symptoms of runny nose due to allergies/cold or other reason
* Current restricted fluid intake for any reason
* Heart disease
* Hypertension
* History of myocardial infarction
* History of cardiac arrhythmia
* Kidney or liver disease
* Vascular disease
* Epilepsy
* Migraine
* Asthma
* Nephritis
* Diabetes and other endocrine diseases
* Frequent or unexplained fainting
* History of stroke
* Aneurysm or brain hemorrhage
* Active psychiatric diagnosis
* Current psychopharmacologic treatment
* Drug or alcohol abuse
* Medical or neurological illness
* Regular use of medication (e.g., vasoconstrictive medications)
* Medication intake less than 2 weeks prior to study (5 weeks for fluoxetine) including daily non-steroidal anti-inflammatory drugs
* Smoking more than 15 cigarettes a day
* Consumption of any alcoholic beverages in the past 24 hours will be excluded
* Elevated blood pressure (>130/90)
* Low blood pressure (<90/60)
* Body temperature >100.1 F

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Speed in social working memory task | Between 40-90 minutes post administration
  Between group differences in the amount of time it takes to perform tasks involving social working memory
Accuracy of deception detection based on self-report | Between 40-90 minutes post administration
  Between group differences in deception detection accuracy based on self-reported ratings of unfamiliar others
Self-reported perceptions of trust and threat | Between 40-90 minutes post administration
  Between group differences in self-reported perceptions of trust and threat towards unfamiliar faces which appear to vary in interpersonal distance
Self-reported empathy and altruistic behavior | Between 40-90 minutes post administration
  Between group differences in self-reported empathy (empathic concern and personal distress), and altruistic behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi I Eisenberger, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Department of Psychology, Los Angeles, California, United States

REFERENCES:
- [Derived] Tabak BA, Teed AR, Castle E, Dutcher JM, Meyer ML, Bryan R, Irwin MR, Lieberman MD, Eisenberger NI. Null results of oxytocin and vasopressin administration across a range of social cognitive and behavioral paradigms: Evidence from a randomized controlled trial. Psychoneuroendocrinology. 2019 Sep;107:124-132. doi: 10.1016/j.psyneuen.2019.04.019. Epub 2019 Apr 29. PMID 31128568
- [Derived] Tabak BA, Meyer ML, Dutcher JM, Castle E, Irwin MR, Lieberman MD, Eisenberger NI. Oxytocin, but not vasopressin, impairs social cognitive ability among individuals with higher levels of social anxiety: a randomized controlled trial. Soc Cogn Affect Neurosci. 2016 Aug;11(8):1272-9. doi: 10.1093/scan/nsw041. Epub 2016 Apr 6. PMID 27053769
- [Derived] Tabak BA, Meyer ML, Castle E, Dutcher JM, Irwin MR, Han JH, Lieberman MD, Eisenberger NI. Vasopressin, but not oxytocin, increases empathic concern among individuals who received higher levels of paternal warmth: A randomized controlled trial. Psychoneuroendocrinology. 2015 Jan;51:253-61. doi: 10.1016/j.psyneuen.2014.10.006. Epub 2014 Oct 17. PMID 25462898